CLINICAL TRIAL: NCT03697967
Title: Supine vs Prone Position During Delayed Cord Clamping in Term Infants A Randomized Trial
Brief Title: Supine vs Prone Position During Delayed Cord Clamping
Acronym: DCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Dr Brahim Bensouda, MD, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-1594
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Newborn; Anemia; Umbilical Cord Problem
Keywords: Delayed cord clamping
MeSH Terms: conditions — Anemia, Neonatal | interventions — Supine Position; Prone Position

STUDY DESIGN:
Intervention Model Description: Randomised two arms study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine (Experimental): Infant placed supine for 120 seconds before cord clamping
  Interventions: Procedure: supine or prone position
- Prone (Experimental): Infant placed prone for 120 seconds before cord clamping
  Interventions: Procedure: supine or prone position

INTERVENTIONS:
Procedure: supine or prone position — Before delivery, a sealed enveloppe is opened by the physician or nurse present at delivery. Immediately at birth the team in charge of delivery place the newborn in skin to skin contact on the mother's chest where he is dried. Umbilical cord clamping is delayed in both intervention arms to 1 minute after birth.
  The newborn is placed in the prone or in the supine position depending on allocation. The nurse in charge of the newborn uses a stopwatch to check the time at which clamping was accomplished.
  All subsequent nursery care are conducted according to hospital protocol.
  Other Names: delay cord clamping

SUMMARY:
This study is conducted to evaluate if the prone position of the newborn on the chest of his mother at birth before delayed cord clamping leads to better hematocrit and hemoglobin at 24-48 hours of life compared to supine position.

DETAILED DESCRIPTION:
At 30 hours of life, laboratory personnel drew a capillary sample from the infant's heel for hemoglobin, hematocrit, and total serum bilirubin at the same time as the newborn metabolic screening sample. There is no added heelstick to routine care, as current standard in our institution requires the bilirubin to be drawn at 30 hours of life.

During universal screening for congenital cardiac defects (30 hours of life), a value of cerebral saturation (CrSO2) is measured using NIRS with INVOS (In Vivo Optical Spectroscopy, INVOS System, Covidien, Dublin, Ireland, Somanetics). Sensors are placed over the forehead and the newborn is in supine position.

ELIGIBILITY:
Inclusion Criteria:

Newborn ≥ 36 weeks gestational age and Born vaginally and Well appearing

Exclusion Criteria:

Out born infant, Infant born by caesarian section, Preterm born less than 36 weeks GA, Infant with intra uterine growth restriction (IUGR: less than 10th percentile) Asphyxiated infant Infant needing immediate resuscitation, Newborn with malformation (gastroschisis, omphalocele, anal atresia, severe head skin injury, congenital cardiac disease Newborn with mother with preeclampsia or gestational hypertension or diabetes on insuline or hemolytic disease or on chemotherapy or on cortisone.

Ages: 1 Minute to 2 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin and hematocrit | 24-48 hours
  Hemoglobin value

SECONDARY OUTCOMES:
Cerebral saturation by near infrared spectroscopy (NIRS) | 24-48 H of life
  Cerebral saturation by near infrared spectroscopy
Bilirubin | 24-48 hours
  Bilirubin value

CONTACTS AND LOCATIONS:
Locations (1):
- Brahim Bensouda, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No